CLINICAL TRIAL: NCT00695539
Title: A Multi-centre, Open Label, Non-randomised, Non Interventional, 24 Weeks Study for the Efficacy and Safety of Rosuvastatin Following Its Administration in Real Life Clinical Practice in Greek Hypercholesterolaemic Patients
Brief Title: Rosuvastatin Efficacy and Safety Evaluation in Hypercholesterolaemic Patients
Acronym: RESEARCH
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Panagiotis Pontikis, MD, Medical & Regulatory Affairs Director, AstraZeneca Greece, AstraZeneca S.A., Greece
Other Study IDs: NIS-CGR-CRE-2007/1
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2009-10-05 (Estimated); Status verified 2009-10

CONDITIONS: Hypercholesterolaemia
Keywords: Rosuvastatin; hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a single-arm, phase IV, open-label, prospective, non interventional study to evaluate the efficacy, tolerability and safety of rosuvastatin administered for 24 weeks in approximately 900 Greek subjects with hypercholesterolemia under normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypercholesterolaemia who are already in treatment with rosuvastatin according to the approved SPC for no longer than 1 month prior to study entry
* Patients that are able to read, understand and sign the Patient Information & Consent Form
* Patients that are willing to comply with all study requirements

Exclusion Criteria:

* Patients that are likely not to comply with all study requirements
* Patients that currently participate or have participated in a 3 months period prior to study entry in another clinical trial
* Female of child bearing potential that do not use a reliable method of contraception. Pregnancy or lactation.
* Patients that meet any of the contraindications described in the approved SPC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care
Sampling Method: Non-Probability Sample
Enrollment: 810 (Actual)
Dates: Start 2007-12; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The assessment of rosuvastatin efficacy in the reduction of low-density lipoprotein cholesterol (LDL-C) in subjects with hypercholesterolemia at week 12 of treatment compared with baseline | At 12 weeks of treatment
To evaluate the percentage of patients on European LDL-C target at week 12 | At 12 weeks of treatment

SECONDARY OUTCOMES:
Changes in HDL-C, TC and TG | At week 12 & 24 of treatment
Safety and tolerability | Throughout the study

CONTACTS AND LOCATIONS:
Locations (6):
- Greece (6):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Iraklio, Crete
  - Research Site, Larissa
  - Research Site, Rio, Patra
  - Research Site, Thessaloniki